CLINICAL TRIAL: NCT04355182
Title: Is Standard 3-degree of External Rotation for Posterior Femoral Cut Relevant for Turkish Population: An Anthropometric MRI Study
Brief Title: Is Standard 3-degree of External Rotation for Posterior Femoral Cut Relevant for Turkish Population
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Nurdan Güngören, Intorn Doctor, Faculty of Medicine, Principal Investigator, Bezmialem Vakif University
Other Study IDs: 3586
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Healthy
Keywords: posterior condylar angle; total knee arthroplasty; external rotation; anthropometric measurements; 3 degrees; Turkish population

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate the posterior condylar angle of the distal femur in Turkish population and its concordance with the current standard prosthesis designs used in total knee arthroplasty and to evaluate anthropometric features of the distal femur in the Turkish population.

DETAILED DESCRIPTION:
The investigators would like to measure condylar twist angles(CTA), posterior condylar angles(PCA), femoral mediolateral lengths (fML), medial femoral anteroposterior lengths(fMAP), lateral femoral anteroposterior lengths (fLAP), distances between trochlear groove and fMAP(DBTG-fMAP), distances between trochlear groove and fLAP(DBTG-fLAP), medial and lateral posterior condylar cartilage thicknesses(MPCCT/LPCCT) on the Magnetic Resonance Images (MRI) of 240 knees of 120 Turkish subjects.

ELIGIBILITY:
Inclusion Criteria:

* non-arthritic knees,

Exclusion Criteria: Patients with,

* intra- or extraarticular deformity on the X-rays or MRIs,
* history of previous extremity surgery,
* history of any systemic disease,
* a BMI of 35 or over.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healty subjects with Turkish ethnic orijin
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-04-12 (Actual)

PRIMARY OUTCOMES:
condylar twist angle and posterior condylar angle | about 5 days
  The condylar twist angle (CTA) is an angle between anatomical transepicondylar axis (TEA),which lying from medial epicondyle to lateral epicondyle of the distal femur, and posterior condylar axis (PCAx). The posterior condylar angle (PCA) is an angle between surgical TEA, which lying from medial epicondylar sulcus to lateral epicondyle, and PCAx[1].

SECONDARY OUTCOMES:
mediolateral lenght of the distal femur (fML) | about 5 days
  The widest mediolateral lenght of the distal femur (fML) in the axial plane which equal to transepicondylar axis
medial anteroposterior lengt (fMAP) and lateral anteroposterior lengt (fLAP) | about 5 days
  the longest anteropesterior distances of the medial and lateral condyles over the cartilage tissue od the distal femur on the axial images[2].
Distance between trochlear groove and fMAP (DBTG-fMAP) and distance between trochlear groove and lateral fAP(DBTG- fLAP) | about 5 days
  MRI sections obtained 3 cm above the tibiofemoral joint will use for evaluation of deepest point of the trochlear groove.The distance between trochlear groove to fMAP and fLAP
Medial and lateral posterior condylar cartilage thicknesses (MPCCT/LPCCT) | about 5 day
  MPCCT/LPCCT were measured at the deepest point in the axial plan.

CONTACTS AND LOCATIONS:
Overall Officials: Nurdan Güngören, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakıf University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Loures FB, Furtado Neto S, Pinto Rde L, Kinder A, Labronici PJ, Goes RF, Marchiori E. Rotational assessment of distal femur and its relevance in total knee arthroplasty: analysis by magnetic resonance imaging. Radiol Bras. 2015 Sep-Oct;48(5):282-6. doi: 10.1590/0100-3984.2014.0037. PMID 26543278
- [Background] Kim TK, Phillips M, Bhandari M, Watson J, Malhotra R. Erratum to: What Differences in Morphologic Features of the Knee Exist Among Patients of Various Races? A Systematic Review. Clin Orthop Relat Res. 2017 May;475(5):1507. doi: 10.1007/s11999-017-5301-1. No abstract available. PMID 28255946